CLINICAL TRIAL: NCT00385580
Title: Phase II Study of Dasatinib (BMS-354825) for Androgen-deprived Progressive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-085
Record Dates: First submitted 2006-10-04; First posted 2006-10-09 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: dasatinib
- 2 (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Tablets, Oral, 100 mg or 70 mg, twice daily, treatment may continue until disease progression
  Other Names: Sprycel; BMS-354825
  Arms: 1
Drug: dasatinib — Tablets, Oral, 100 mg, once daily (QD) treatment may continue until disease progression
  Arms: 2

SUMMARY:
The purpose of this study is to learn if men with metastatic prostate cancer and rising Prostate Specific Antigen (PSA), who have been surgically castrated or are undergoing androgen deprivation with Luteinizing Hormone Releasing Hormone (LHRH) treatment, respond to dasatinib. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* males, 18 or older
* proven advanced prostate cancer
* documented metastatic disease
* rising PSA levels
* castrate levels of testosterone

Exclusion Criteria:

* symptomatic CNS (brain or spinal cord) metastasis
* medical condition which may increase the risk of toxicity
* any prior or ongoing anti-cancer medical therapy or immunotherapy for prostate cancer other than primary androgen deprivation agents
* unable to take oral medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (7):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University Of Chicago, Chicago, Illinois
  - The Bunting Blaustein Cancer Research Building, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center-Sidney Kimmel Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University Of Wisconsin Paul P Carbone Comprehensive Ca Ctr, Madison, Wisconsin
- France (3):
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Villejuif
- Local Institution, Rome, Italy

REFERENCES:
- [Background] Yu EY, Wilding G, Posadas E, Gross M, Culine S, Massard C, Morris MJ, Hudes G, Calabro F, Cheng S, Trudel GC, Paliwal P, Sternberg CN. Phase II study of dasatinib in patients with metastatic castration-resistant prostate cancer. Clin Cancer Res. 2009 Dec 1;15(23):7421-8. doi: 10.1158/1078-0432.CCR-09-1691. Epub 2009 Nov 17. PMID 19920114
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 130 participants were enrolled in the study; 95 participants entered the treatment period. 67 discontinued due to disease progression, 13 for study drug toxicity, 5 for other reasons, 4 withdrew consent, 2 for adverse events unrelated to the study, 2 requested discontinuation, 1 due to death, and 1 due to maximum clinical benefit.
Groups:
- Dasatinib 100 mg Once Daily (QD): Participants were administered an oral dose of 100 mg dasatinib tablet QD. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 100 mg or 70 mg Twice Daily (BID): Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 200 mg which was later decreased to 70 mg BID for a TDD of 140 mg. Of the 47 treated participants in the BID group, 25 received 100 mg and 22 received 70 mg of dasatinib as their starting doses. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Period: Overall Study
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Started | 48 (Number of participants treated.) | 47 (Number of participants treated.)
Completed | 48 (Completed=off study. Major reasons for being off study are disease progression, and study toxicity.) | 47 (Completed=off study. Major reasons for being off study are disease progression, and study toxicity.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID) | Total
Number analyzed (Participants) | 48 | 47 | 95
Age Continuous [Median (Full Range); unit: years] | 68.0 [47.0 to 85.0] | 70.0 [54.0 to 87.0] | 69.0 [47.0 to 87.0]
Age, Customized [Number; unit: participants]
  < 65 years | 12 | 13 | 25
  >=65 years | 36 | 34 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 48 | 47 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 15 | 16 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 46 | 45 | 91
  Black/African American | 1 | 2 | 3
  Hispanic | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG)Performance Status (PS) [Number; unit: participants] — The ECOG PS is used to assess disease severity. A score of 0 is normal activity; 1 is symptoms, but fully ambulatory; 2 is symptomatic, but in bed < 50% of the day; 3 is needs to be in bed > 50% of the day, but not bedridden; 4 is unable to get out of bed; 5 is dead.
  participants
    0=normal activity | 35 | 28 | 63
    1=symptoms, but fully ambulatory | 13 | 18 | 31
    2=symptomatic, but in bed < 50% of the day. | 0 | 1 | 1
    3=needs to be in bed >50% of day, not bedridden | 0 | 0 | 0
    4=unable to get out of bed | 0 | 0 | 0
    5=dead | 0 | 0 | 0
Height continuous [Mean (Standard Deviation); unit: centimeter (cm)] | 174.44 (7.35) | 172.63 (12.67) | 173.58 (10.19)
Weight continuous [Mean (Standard Deviation); unit: kilogram (Kg)] | 92.50 (18.25) | 89.16 (14.72) | 90.85 (16.60)
FACT Advanced Prostate Symptom Index (FAPSI) -8 Score from baseline [Median (Full Range); unit: Units on a scale] — FAPSI-8:symptom index of important clinician-rated symptoms/concerns to monitor when assessing value of treatment for advanced prostate cancer. Participants respond to each item on a 5-point Likert-type scale from 0 (not at all) to 4 (very much). GP1:I have lack of energy, GP4:I have pain, GE6:I worry that my condition will get worse, C2: I am losing weight, P2:I have certain areas in my body where I experience significant pain,P3:My pain keeps me from doing things I want to do, P7:I have difficulty urinating, P8:My problems with urinating limit my activities.
  Units on a scale
    Total Score | 26.00 [15.00 to 31.00] | 26.00 [13.00 to 31.00] | 26.00 [15.00 to 31.00]
    GP1 | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00]
    GP4 | 3.00 [1.00 to 4.00] | 3.00 [1.00 to 4.00] | 3.00 [1.00 to 4.00]
    GE6 | 3.00 [0.00 to 4.00] | 2.00 [0.00 to 4.00] | 2.00 [0.00 to 4.00]
    C2 | 4.00 [0.00 to 4.00] | 4.00 [2.00 to 4.00] | 4.00 [0.00 to 4.00]
    P2 | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00]
    P3 | 4.00 [0.00 to 4.00] | 4.00 [1.00 to 4.00] | 4.00 [0.00 to 4.00]
    P7 | 4.00 [0.00 to 4.00] | 4.00 [0.00 to 4.00] | 4.00 [0.00 to 4.00]
    P8 | 4.00 [0.00 to 4.00] | 4.00 [1.00 to 4.00] | 4.00 [0.00 to 4.00]
Urinary N-telopeptide (uNTx)Value from Baseline [Number; unit: Participants] — uNTx is a measure of bone metabolism decrease in the marker relative to baseline indicates a decrease in bone metabolism.
  Participants
    < 60 nanomol (nmol)/mmol creatinine | 26 [10.0 to 89.0] | 28 [4.0 to 86.0] | 54
    >= 60 nmol/mmol creatinine | 20 | 15 | 35
    Unknown uNTx value | 2 | 4 | 6
Bone-specific Alkaline Phosphatase (BAP) Value from baseline [Number; unit: Participants] — BAP is a measure of bone metabolism. A decrease in BAP relative to baseline indicates a decrease in bone metabolism.
  Participants
    High >41.3 U/L | 18 [6.0 to 88.0] | 19 [4.0 to 62.0] | 37
    Low <15 U/L | 3 | 2 | 5
    Normal 15-41.3 U/L | 26 | 22 | 48
    Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response = confirmed prostate specific antigen (PSA) response (decrease in PSA =>50% from baseline), confirmed improved bone scan (disappearance of => 1 lesion, no new lesions, new pain not developing), confirmed complete response (CR: disappearance of all lesions) or confirmed partial response (PR: =>30% in sum of longest diameter [LD] of all lesions compared to baseline sum LD), stable disease (SD: neither sufficient increase for progressive disease [PD: =>20% increase in sum of LD of all target lesions] nor sufficient shrinkage for PR), based on Response Criteria in Solid Tumors [RECIST].
Time Frame: Within 2 weeks of first study drug administration, thereafter recorded every 4 weeks.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants | 12 | 13

2. Primary Outcome: Percentage of Participants With a Response
Description: Response = confirmed PSA response (decrease in PSA =>50% from baseline), confirmed improved bone scan (disappearance of => 1 lesion, no new lesions, new pain not developing), confirmed CR (disappearance of all lesions) or confirmed PR (=>30% in sum of LD of all lesions compared to baseline sum LD), SD (neither sufficient increase for PD [=>20% increase in sum of LD of all target lesions] nor sufficient shrinkage for PR), based on RECIST.
Time Frame: Within 2 weeks of first study drug administration, thereafter recorded every 4 weeks.
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
Percentage of Participants | 25.00 [13.64 to 39.60] | 27.70 [15.62 to 42.64]

3. Secondary Outcome: Number of Participants With a Decrease in PSA by at Least 50% From Baseline
Description: PSA is a marker of prostate cancer and a PSA response is defined as a decrease in the PSA value by at least 50% from baseline, for 2 successive evaluations, each at least 2 weeks apart, for a total of 3 measurements.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All PSA response-evaluable participants: participants who had pre-treatment PSA measurements and at least 2 on-study PSA measurements.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 43 | 43
participants | 1 | 1

4. Secondary Outcome: Percentage of Participants With a Decrease in PSA by at Least 50% From Baseline
Description: PSA is a marker of prostate cancer and a PSA response is defined as a decrease in the PSA value by at least 50% from baseline for 2 successive evaluations, each at least 2 weeks apart, for a total of 3 measurements.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 43 | 43
Percentage of Participants | 2.3 | 2.3

5. Secondary Outcome: Number of Months of Decrease in PSA by at Least 50% From Baseline
Description: PSA is a marker of prostate cancer. The duration of PSA response is measured from the time that the first of the 2 consecutive measurements met the criteria for confirmed PSA response, until the date of the first of the 3 consecutive measurements that confirm PSA progression, or the date of disease progression, or the date of death.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: Participants with a decrease in PSA by at least 50% from baseline
Measure: Number; unit: months
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 1 | 1
months | 0.82 | 11.17

6. Secondary Outcome: Number of Participants With Decrease in PSA Velocity
Description: PSA is a marker of prostate cancer. PSA velocity measures the rate of change of PSA values. A decrease in PSA values and hence PSA velocity is an early indicator of potential anti-tumor activity.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All PSA response-evaluable participants: participants who had 2 or more pre-treatment PSA measurements and at least 2 on-study PSA measurements.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 43 | 43
participants | 25 [-0.4 to 5.7] | 16 [-0.2 to 13.2]

7. Secondary Outcome: Number of Participants With Decrease in PSA Log Slope
Description: PSA is a marker of prostate cancer. A decrease in PSA value is an early indicator of potential anti-tumor activity. Log (PSA) is assumed to have a linear relationship with time. The PSA log slope is defined as the slope of the log PSA line.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 43 | 43
participants | 38 [-0.015 to 0.018] | 34 [-0.008 to 0.029]

8. Secondary Outcome: Number of Participants With Increase in PSA Doubling Time
Description: PSA is a marker of prostate cancer. PSA doubling time is defined as log 2 divided by the slope of the log PSA line. An increase in PSA doubling time indicates improvement in anti-tumor activity.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All PSA response-evaluable participants: participants who had 2 or more pre-treatment PSA measurements and at least 2 on-study PSA measurements and positive log slope pre-treatment and on-study measurements.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 38 | 41
participants | 34 [39.0 to 858.0] | 32 [24.0 to 2622.0]

9. Secondary Outcome: Number of Participants With CR or PR
Description: Tumor response was defined as the number of participants whose best response was CR or PR, per RECIST: CR: disappearance of all target/non-target lesions; PR: >= 30% decrease in the sum of the LDs of target lesions relative to the baseline sum LD
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All response-evaluable participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 18 | 21
participants | 1 | 0

10. Secondary Outcome: Number of Participants With CR, PR or SD
Description: Disease control rate is defined as the number of participants whose best response was CR, PR or SD, per RECIST: CR: disappearance of all target/non-target lesions; PR: >= 30% decrease in the sum of the LDs of target lesions relative to the baseline sum LD; SD: neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR; PD: defined as appearance of new lesion/s, or >=20% increase in the sum of the LD of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All response-evaluable participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 18 | 21
participants | 11 | 12

11. Secondary Outcome: Number of Participants With a Confirmed Improved Bone Scan
Description: An improved bone scan was defined as 1 or more of the following: disappearance of at least 1 lesion, no new lesions appearing since the most recent prior assessment, or new pain not developing in an area that was previously visualized. A response is considered confirmed if it is noted on 2 examinations at least 4 weeks apart.
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All response-evaluable participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 40 | 38
participants | 0 | 1

12. Secondary Outcome: Percentage of Participants With Confirmed Improved Bone Scan
Description: as for outcome 11
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: Participants with confirmed improved bone scan.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 40 | 38
Percentage of Participants | 0.0 | 2.6

13. Secondary Outcome: Number of Participants With Disease Progression
Description: Disease progression: progression of target lesions or unequivocal progression of non-measurable lesions/disease as evaluated by computed tomography (CT) scan or magnetic resonance imaging (MRI), not as evaluated by bone scan (non-measurable lesions included visceral and bone lesions), loss of PSA response (only for participants who achieved a PSA response) or Investigator-defined clinical progression based on physical examination, history, symptoms, and ECOG-PS. For participants who did not progress or die, date of last PSA measurement or tumor assessment was used, whichever occurred first.
Time Frame: Prior to treatment with the study drug, Week 12 and every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants | 30 | 34

14. Secondary Outcome: Median Number of Months to Disease Progression
Description: Measured from date of first dose to date of first 3 consecutive measurements that confirm PSA progression, date of disease progression,or death date.Disease progression:progression of target lesions or unequivocal progression of non-measurable lesions/disease as evaluated by computed tomography (CT) scan or magnetic resonance imaging (MRI),loss of PSA response or Investigator-defined clinical progression based on physical examination,history,symptoms,and ECOG-PS.For participants who did not progress or die,date of last PSA measurement or tumor assessment was used, whichever occurred first.
Time Frame: Prior to treatment with the study drug, Week 12 and every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
months | 4.7 [2.8 to 5.5] | 2.8 [2.8 to 5.4]

15. Secondary Outcome: Median Change From Baseline in Individual FAPSI Scores at Week 12
Description: FAPSI-8:symptom index of important clinician-rated symptoms/concerns to monitor when assessing value of treatment for advanced prostate cancer. Participants respond to each item on a 5-point Likert-type scale from 0 (not at all) to 4 (very much). GP1:I have lack of energy, GP4:I have pain, GE6:I worry that my condition will get worse, C2: I am losing weight, P2:I have certain areas in my body where I experience significant pain,P3:My pain keeps me from doing things I want to do, P7:I have difficulty urinating, P8:My problems with urinating limit my activities.
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
Units on a scale
  GP1 | 0.00 [-2.00 to 2.00] | -1.00 [-4.00 to 3.00]
  GP4 | 0.00 [-2.00 to 2.00] | 0.00 [-2.00 to 2.00]
  GE6 | 0.00 [-3.00 to 2.00] | 0.00 [-2.00 to 3.00]
  C2 | 0.00 [-3.00 to 3.00] | 0.00 [-3.00 to 1.00]
  P2 | 0.00 [-3.00 to 1.00] | 0.00 [-2.00 to 2.00]
  P3 | 0.00 [-1.00 to 2.00] | 0.00 [-3.00 to 3.00]
  P7 | 0.00 [-4.00 to 2.00] | 0.00 [-3.00 to 2.00]
  P8 | 0.00 [-1.00 to 1.00] | 0.00 [-3.00 to 2.00]

16. Secondary Outcome: Median Change From Baseline in Total FAPSI-8 Scores at Weeks 12, 24 and 36
Description: The FAPSI-8 is a symptom index comprised of the most important clinician-rated symptoms or concerns to monitor when assessing the value of treatment for advanced prostate cancer. It includes 8 items developed to measure symptoms/concerns specific to prostate cancer such as fatigue, pain (3-items), weight loss, difficulty with urination (2-items) and concerns about the condition becoming worse. Participants respond to each item on a 5-point Likert-type scale from 0 (not at all) to 4 (very much).
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
Units on a scale
  Week 12 (n=26, 29) | 0.00 [-11.00 to 4.00] | -2.00 [-12.00 to 6.00]
  Week 24 (n=14, 6) | -2.50 [-8.00 to 1.00] | -2.00 [-11.00 to 4.00]
  Week 36 (n=4, 5) | NA [NA to NA] — Week 36 data was not summarized in the CSR because of the small N, and it was agreed that the summaries based on small N were not interpretable. | NA [NA to NA] — Week 36 data was not summarized in the CSR because of the small N, and it was agreed that the summaries based on small N were not interpretable.

17. Secondary Outcome: Median Change From Baseline in Individual FAPSI Scores at Week 24
Description: as for outcome 15
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
Units on a scale
  GP1 | 0.00 [-2.00 to 1.00] | 0.00 [-2.00 to 0.00]
  GP4 | -0.50 [-3.00 to 0.00] | -0.50 [-1.00 to 2.00]
  GE6 | -0.50 [-2.00 to 2.00] | -0.50 [-1.00 to 1.00]
  C2 | 0.00 [-2.00 to 3.00] | -0.50 [-2.00 to 0.00]
  P2 | 0.00 [-2.00 to 1.00] | 0.00 [-3.00 to 1.00]
  P3 | 0.00 [-1.00 to 1.00] | 0.00 [-4.00 to 1.00]
  P7 | 0.00 [-2.00 to 1.00] | 0.00 [-1.00 to 0.00]
  P8 | 0.00 [-2.00 to 1.00] | 0.00 [0.00 to 0.00]

18. Secondary Outcome: Median Change From Baseline in Individual FAPSI Scores at Week 36
Description: FAPSI-8:index of symptoms/concerns when assessing value of treatment for advanced prostate cancer.Participants respond to each item on 5-point Likert-type scale:0 (not at all) to 4 (very much).GP1:I have lack of energy,GP4:I have pain,GE6:I worry that my condition will get worse,C2:I am losing weight,P2:I have certain areas in my body where I experience significant pain,P3:My pain keeps me from doing things I want to do,P7:I have difficulty urinating,P8:My problems with urinating limit my activities. The number of participants for whom these data are available is too small for analysis.
Time Frame: Prior to treatment with the study drug, Week 12, every 12 weeks thereafter and at the end of the treatment.
Population: All treated participants. The number of participants for whom this data are available is too small for analysis.
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs) or Discontinuations Due to AEs
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Deaths | 2 | 2
  AEs | 48 | 47
  SAEs | 10 | 11
  All AEs Leading to Discontinuation | 13 | 8

20. Secondary Outcome: Number of Participants Who Experienced Drug-related SAEs, Drug-related AEs, Drug-related Grade 3/4 AEs and Discontinuations Due to Drug-related AEs.
Description: Drug-related AEs are those events with a relationship to the study therapy of certain; probable; possible; or missing. Drug-related SAEs are those events with any relationship to the study therapy. Drug-related AEs were graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 3.0: Grade 1=mild, 2=moderate, 3=severe, 4=life threatening, 5=death. Participants who discontinued the study due to any drug-related AEs were also recorded.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Drug-related SAEs | 1 | 6
  Drug-related AEs | 43 | 47
  Drug-related Grade 3-4 AEs | 7 | 15
  Drug-related AEs Leading to Discontinuation | 9 | 7

21. Secondary Outcome: Number of Participants With Grade 3-4 Hematology Abnormalities
Description: Abnormalities were graded per the NCI CTC, version 3.0 criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: Hemoglobin: Grade 3:6.5 - <8.0g/dL, Grade 4: <6.5g/dL. Platelets: Grade 3: 25.0 - <50.0*10^9/L, Grade 4: <25.0*10. Absolute Neutrophil Count (ANC): Grade 3: 0.5 - <1.0*10^9/L, Grade 4: <0.5*10^9/L. Leukocytes: Grade 3: 1.0 - <2.0*10^9/L, Grade 4: <1.0*10^9/L.
Time Frame: Data was collected prior treatment with the study drug, Week 2, Week 4, Week 8, Week 12 , every 4 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Absolute Neutrophil Count (ANC) | 0 | 1
  Hemoglobin | 0 | 1
  Platelet Count | 0 | 1
  Leukocytes | 0 | 0

22. Secondary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities in Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Bilirubin and Calcium
Description: Abnormalities were graded according to the NCI CTC, version 3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase: Grade 3: 5.0-20.0 * ULN (upper limit of normal), Grade 4: >20.0 * ULN; calcium: Grade 3: 6.0-<7.0 or >12.5-13.5 mg/dL, Grade 4: <0.6->13.5 mg/dL; bilirubin: Grade 3: >3-10 * ULN, Grade 4: >10 * ULN.
Time Frame: as for outcome 21
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Alanine Aminotransferase | 0 | 0
  Aspartate Aminotransferase | 0 | 0
  Alkaline Phosphatase | 6 | 0
  Bilirubin | 0 | 0
  Hypercalcemia | 0 | 0
  Hypocalcemia | 1 | 0

23. Secondary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities in Creatinine, Potassium, Sodium and Phosphorous
Description: Abnormalities were graded per the NCI CTC, version 3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: phosphorous: Grade 3: 1.0-<2.0 mg/dL, Grade 4: <1.0 mg/dL; sodium: Grade 3: 120-<130 or >155-160mEq/L, Grade 4: <120 or >160 mEq/L; creatinine: Grade 3: >3.0-6.0 * ULN, Grade 4: >6.0 * ULN; potassium: Grade 3: 2.5 -<3.0 or >6.0 -7.0 mEq/L, Grade 4: < 2.5 or >7.0 mEq/L.
Time Frame: as for outcome 21
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Creatinine | 0 | 0
  Hyperkalemia | 0 | 0
  Hypokalemia | 2 | 1
  Hypernatremia | 0 | 0
  Hyponatremia | 1 | 1
  Phosphorus, Inorganic | 2 | 2

24. Secondary Outcome: Number of Participants With Abnormal Lactate Dehydrogenase (LD)
Description: LDH is a laboratory safety parameter. Normal ranges for LD vary with both age and disease status, and another reason for variation in upper limit of normal (ULN) and lower limit of normal (LLN) is that LD was measured via a local (versus a standardized) laboratory. It is therefore not possible to provide one ULN and LLN for the population.
Time Frame: Data was collected prior treatment with the study drug, Week 2, Week 4, Week 8, Week 12, every 4 weeks thereafter and at the end of the treatment.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants | 33 | 41

25. Secondary Outcome: Number of Participants With Positive Urinalysis
Description: Participants' urine samples were tested for the presence of blood, glucose and protein. If these substances were present in a participant's urine, the results were given as "positive".
Time Frame: as for outcome 21
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants
  Blood | 20 | 21
  Glucose | 2 | 1
  Protein | 21 | 26

26. Secondary Outcome: Number of Participants With QTc Prolongation
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTc is the QT interval corrected for heart rate. A prolonged QT interval is a risk factor for ventricular tachyarrhythmias and sudden death.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 48 | 47
participants | 3 | 10

27. Secondary Outcome: Number of Participants With a Baseline uNTx Value <=ULN, With a Decrease, Increase or no Change in uNTx
Description: uNTx is a measure of bone metabolism. A decrease in the marker relative to baseline indicates a decrease in bone metabolism.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All treated participants who had a baseline uNTx value <=ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 26 | 26
participants
  0-35 percent decrease | 2 | 6
  >35-70 percent decrease | 13 | 12
  >70 percent decrease | 5 | 1
  No change or increase | 6 | 7

28. Secondary Outcome: Number of Participants With a Baseline uNTx Value >ULN, With a Decrease, Increase or no Change in uNTx
Description: as for outcome 27
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All treated participants who had a baseline uNTx value >ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 17 | 15
participants
  0-35 percent decrease | 6 | 4
  >35-70 percent decrease | 3 | 9
  >70 percent decrease | 4 | 1
  No change or increase | 4 | 1

29. Secondary Outcome: Number of Participants With a uNTx Response
Description: uNTx is a measure of bone metabolism. uNTx response is defined for participants with baseline uNTx above ULN. It is defined as either on-study uNTx values decreasing to within normal limits or 35% or more decrease in uNTx from baseline, whichever happens first.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: Participants with a baseline uNTx value > ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 17 | 15
participants | 10 | 10

30. Secondary Outcome: Median Number of Months of uNTx Response
Description: uNTx is a measure of bone metabolism.The median number of months of uNTx response was calculated for participants with baseline uNTx =< ULN and uNTx progression during treatment, from first dose of dasatinib to uNTx progression.For participant with baseline uNTx above ULN, it was time from uNTx response to uNTx progression.For participants with baseline uNTx equal to or below ULN or uNTx response and no uNTx progression, the date of last uNTx assessment was used. Duration of uNTx response was not defined for participants with baseline value greater than ULN who never achieved uNTx responses.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: Participants who demonstrated a uNTx response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 10 | 10
months | NA [6.3 to NA] — Not enough participants with response had progressed; therefore, median and upper limit of 95% confidence interval could not be estimated. | NA [4.7 to NA] — Not enough participants with response had progressed; therefore, median and upper limit of 95% confidence interval could not be estimated.

31. Secondary Outcome: Number of Participants With a Baseline BAP Value <= ULN, With a Decrease, Increase or no Change in BAP
Description: BAP is a measure of bone metabolism. A decrease in BAP relative to the baseline indicates decrease in bone metabolism.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All treated participants who had a baseline BAP value <=ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 28 | 23
participants
  0-35 percent decrease | 12 | 14
  >35-70 percent decrease | 5 | 2
  >70 percent decrease | 1 | 0
  No change or increase | 10 | 7

32. Secondary Outcome: Number of Participants With a Baseline BAP Value > ULN, With a Decrease, Increase or no Change in BAP
Description: BAP is a measure of bone metabolism. A decrease in BAP relative to baseline indicates a decrease in bone metabolism.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: All treated participants who had a baseline BAP value >ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 16 | 17
participants
  0-35 percent decrease | 6 | 6
  >35-70 percent decrease | 1 | 3
  >70 percent decrease | 1 | 0
  No change or increase | 8 | 8

33. Secondary Outcome: Number of Participants With BAP Response
Description: BAP is a measure of bone metabolism. A BAP response is calculated for participants with a baseline BAP value > ULN. It is defined as on-study BAP values within normal limits.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: Participants with a baseline BAP value > ULN and at least 1 on-study value.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 16 | 17
participants | 4 | 5

34. Secondary Outcome: Median Number of Months of BAP Response
Description: The median number of months of the BAP response was calculated for participants with baseline BAP <= ULN, from first dose of dasatinib to the first time BAP is above ULN. For participants with baseline BAP > ULN, it was the time from BAP response to the first time BAP was above ULN. For participants with baseline BAP =< ULN or BAP, and no BAP above ULN, last BAP assessment date was used. The median number of months of response was not defined for participants with baseline value > ULN, that never achieved BAP response.
Time Frame: Prior to treatment with the study drug, Week 4, Week 8, Week 12 and every 4 weeks thereafter.
Population: Participants who demonstrated a BAP response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg or 70 mg Twice Daily (BID)
Number analyzed (Participants) | 4 | 5
months | NA [NA to NA] — Not enough participants with response had progressed; therefore, median and 95% confidence interval could not be estimated. | NA [NA to NA] — Not enough participants with response had progressed; therefore, median and 95% confidence interval could not be estimated.

35. Secondary Outcome: Mean Plasma Concentration at 100 mg Dasatinib Dose (Week 2)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID and QD group.
Population: All available concentration-time data from participants who received at least 1 dose of dasatinib. The 'n' is signifying those who were evaluated for this measure at timepoint for each group respectively. Data are split by actual dose administered. If there was dose modification, participant was grouped according to dose given on PK collection day.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dasatinib 100 mg Once Daily (QD): Participants were administered an oral dose of 100 mg dasatinib tablet QD (100 dose). Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 100 mg Twice Daily (BID): Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 200 mg (100 dose). Of the 47 treated participants in the BID group, 25 received 100 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 70 mg BID: Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 70 mg BID for a TDD of 140 mg (100 dose). Of the 47 treated participants in the BID group, 22 received 70 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 48 | 25 | 22
ng/mL
  0 hour (n=39,18,1) | 3.17 (4.03) | 8.15 (4.53) | 5.46 (0.00)
  1hour (n=41,19,1) | 102.98 (81.80) | 73.05 (64.51) | 83.24 (0.00)
  3 hour (n=41,19,1) | 45.28 (27.06) | 37.58 (25.10) | 23.73 (0.00)
  6 hour (n=41,18,1) | 19.37 (13.77) | 15.02 (7.66) | 8.88 (0.00)
  12 hour (n=30,12,1) | 16.86 (55.72) | 10.51 (8.98) | 9.89 (0.00)

36. Secondary Outcome: Mean Plasma Concentration at 100 mg Dasatinib Dose (Week 6)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID and QD group.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 48 | 25 | 22
ng/mL
  0 hour (n=31,8,1) | 15.46 (72.21) | 10.61 (4.27) | 8.68 (0.00)
  1hour (n=36,9,1) | 89.55 (78.64) | 59.75 (35.86) | 78.78 (0.00)
  3 hour (n=36,9,1) | 40.10 (31.21) | 33.26 (16.74) | 29.85 (0.00)
  6 hour (n=36,9,1) | 15.15 (8.24) | 16.27 (9.18) | 13.68 (0.00)
  12 hour (n=26,8,1) | 17.27 (29.64) | 15.92 (10.34) | 13.93 (0.00)

37. Secondary Outcome: Mean Plasma Concentration at 70 mg Dasatinib Dose (Week 2)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID and QD group.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dasatinib 100 mg Once Daily (QD): Participants were administered an oral dose of 100 mg dasatinib tablet QD (70 dose). Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 100 mg Twice Daily (BID): Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 200 mg (70 dose). Of the 47 treated participants in the BID group, 25 received 100 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 70 mg BID: Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 70 mg BID for a TDD of 140 mg (70 dose). Of the 47 treated participants in the BID group, 22 received 70 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 48 | 25 | 22
ng/mL
  0 hour (n=1,1,17) | 2.16 (0.00) | 11.69 (0.00) | 7.08 (3.76)
  1hour (n=1,1,20) | 140.15 (0.00) | 10.37 (0.00) | 66.47 (43.94)
  3 hour (n=1,1,20) | 43.50 (0.00) | 44.90 (0.00) | 27.60 (13.28)
  6 hour (n=1,1,19) | 17.09 (0.00) | 52.77 (0.00) | 14.01 (6.06)
  12 hour (n=1,1,18) | 24.52 (0.00) | 12.54 (0.00) | 11.91 (15.82)

38. Secondary Outcome: Mean Plasma Concentration at 70 mg Dasatinib Dose (Week 6)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID group.
Population: All available concentration-time data from participants who received at least 1 dose of dasatinib. The 'n' is signifying those who were evaluated for this measure at timepoint for each group respectively. Data are split by actual dose administered. In treatment group (100 mg, QD), no participant received a 70 mg at PK collection day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 0 | 25 | 22
ng/mL
  0 hour (n=9,12) |  | 7.29 (3.76) | 6.05 (3.13)
  1hour (n=10,11) |  | 54.67 (42.75) | 77.83 (55.72)
  3 hour (n=10,12) |  | 30.98 (25.78) | 24.17 (12.34)
  6 hour (n=8,11) |  | 16.13 (9.77) | 11.81 (5.48)
  12 hour (n=5,11) |  | 7.72 (4.24) | 16.29 (31.40)

39. Secondary Outcome: Mean Plasma Concentration at 50 mg Dasatinib Dose (Week 2)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID and QD group.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dasatinib 100 mg Once Daily (QD): Participants were administered an oral dose of 100 mg dasatinib tablet QD (50 dose). Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 100 mg Twice Daily (BID): Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 200 mg (50 dose). Of the 47 treated participants in the BID group, 25 received 100 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 70 mg BID: Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 70 mg BID for a TDD of 140 mg (50 dose). Of the 47 treated participants in the BID group, 22 received 70 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 48 | 25 | 22
ng/mL
  0 hour (n=2,2,1) | 2.28 (0.67) | 7.39 (7.7) | 14.21 (0.00)
  1hour (n=2,2,1) | 60.35 (37.22) | 42.15 (42.53) | 117.71 (0.00)
  3 hour (n=2,2,1) | 28.38 (12.06) | 23.18 (22.22) | 57.08 (0.00)
  6 hour (n=2,2,1) | 12.96 (2.99) | 6.09 (3.92) | 23.63 (0.00)
  12 hour (n=2,2,1) | 47.97 (64.93) | 12.90 (11.13) | 15.92 (0.00)

40. Secondary Outcome: Mean Plasma Concentration at Dose 50 mg (Week 6)
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose, 1 hour, 3 hours, 6 hours and at 12 hours after any dose for BID and QD group.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dasatinib 100 mg Twice Daily (BID): Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 200 mg (X dose). Of the 47 treated participants in the BID group, 25 received 100 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 70 mg BID: Participants were administered an oral dose of 100 mg dasatinib tablet BID for a total daily dose (TDD) of 70 mg BID for a TDD of 140 mg (X dose). Of the 47 treated participants in the BID group, 22 received 70 mg of dasatinib as their starting dose. Participants continued to receive the study drug as long as tolerated or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | Dasatinib 100 mg Once Daily (QD) | Dasatinib 100 mg Twice Daily (BID) | Dasatinib 70 mg BID
Number analyzed (Participants) | 48 | 25 | 22
ng/mL
  0 hour (n=1,1,3) | 3.54 (0.00) | 7.43 (0.00) | 3.68 (1.48)
  1hour (n=1,1,4) | 134.89 (0.00) | 62.62 (0.00) | 31.99 (22.32)
  3 hour (n=1,1,4) | 27.35 (0.00) | 20.65 (0.00) | 13.28 (2.67)
  6 hour (n=1,1,3) | 13.20 (0.00) | 10.29 (0.00) | 7.50 (1.29)
  12 hour (n=1,1,3) | 2.16 (0.00) | 8.33 (0.00) | 3.12 (0.54)

ADVERSE EVENTS:
Groups:
- Dasatinib: All treated participants
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 21/95
Other Adverse Events (participants affected / at risk) | 94/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=95)
HAEMOGLOBIN (Investigations) | 2
PLATELET COUNT (Investigations) | 1
BLOOD PRESSURE DECREASED (Investigations) | 1
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1
ATRIAL FLUTTER (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ISCHAEMIA (Vascular disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SEPSIS (Infections and infestations) | 1
BACTERAEMIA (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
HUMAN EHRLICHIOSIS (Infections and infestations) | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
PYREXIA (General disorders) | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=95)
WEIGHT DECREASED (Investigations) | 13
WEIGHT INCREASED (Investigations) | 7
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 13
ATRIAL FIBRILLATION (Cardiac disorders) | 6
PERICARDIAL EFFUSION (Cardiac disorders) | 12
FLUSHING (Vascular disorders) | 10
HOT FLUSH (Vascular disorders) | 6
DEPRESSION (Psychiatric disorders) | 7
HEADACHE (Nervous system disorders) | 32
DIZZINESS (Nervous system disorders) | 12
DYSGEUSIA (Nervous system disorders) | 6
NAUSEA (Gastrointestinal disorders) | 37
VOMITING (Gastrointestinal disorders) | 14
DIARRHOEA (Gastrointestinal disorders) | 45
FLATULENCE (Gastrointestinal disorders) | 10
CONSTIPATION (Gastrointestinal disorders) | 18
ABDOMINAL PAIN (Gastrointestinal disorders) | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5
RHINITIS (Infections and infestations) | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6
HAEMATURIA (Renal and urinary disorders) | 7
DECREASED APPETITE (Metabolism and nutrition disorders) | 39
ANAEMIA (Blood and lymphatic system disorders) | 10
RASH (Skin and subcutaneous tissue disorders) | 25
ALOPECIA (Skin and subcutaneous tissue disorders) | 5
DRY SKIN (Skin and subcutaneous tissue disorders) | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16
BONE PAIN (Musculoskeletal and connective tissue disorders) | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 17
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 27
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 33
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 8
CHILLS (General disorders) | 5
OEDEMA (General disorders) | 8
FATIGUE (General disorders) | 44
PYREXIA (General disorders) | 17
ASTHENIA (General disorders) | 24
OEDEMA PERIPHERAL (General disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.